CLINICAL TRIAL: NCT03800394
Title: Pharmacokinetics of Anti-tuberculosis and Antiretroviral Drugs in Children
Brief Title: Pharmacokinetics of Intracellular TFV-DP and FTC-TP in HIV-infected Adolescents
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201801820 - PKAdol; 2R01HD071779 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Human Immunodeficiency Virus (HIV); Tuberculosis; Coinfection
Keywords: Pharmacokinetic; Pharmacogenomic; Tenofovir diphosphate; Emtricitabine triphosphate; Adolescents
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral mononuclear cells (PBMCs) and deoxyribonucleic acid (DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- HIV only: Adolescents aged 10-19 years with HIV infection
  Interventions: Other: Observational PK study
- HIV/TB: Adolescents aged 10-19 years with HIV and TB coinfection
  Interventions: Other: Observational PK study

INTERVENTIONS:
Other: Observational PK study — Effect of antituberculosis treatment, age and genetic factors on intracellular TFV-DP and FTC-TP concentrations

SUMMARY:
Tenofovir (TFV) disoproxil fumarate (TDF) plus emtricitabine (FTC) or lamivudine (3TC) is the preferred nucleoside backbone of first-line antiretroviral therapy (ART) for adolescents in sub-Saharan Africa. In addition, TDF/FTC is recommended for preexposure prophylaxis (PrEP) for human immunodeficiency virus (HIV) infection in adolescents at substantial risk of acquisition of HIV infection, as well as for hepatitis B virus (HBV) treatment in those with HBV/HIV coinfection. The efficacy TDF and FTC are dependent on intracellular concentrations of the active phosphate anabolites, called TFV diphosphate (TFV-DP) and FTC triphosphate (FTC-TP). However, the intracellular pharmacokinetics of TFV-DP and FTC-TP to examine the adequacy of current dosages in African adolescents has not been previously studied. Thus, examining the pharmacokinetics (PK) of these widely used antiretrovirals in African adolescents is important as ART outcomes remain poor and the recommended dosages of these drugs for children and adolescent were extrapolated from drug approval clinical trials in adult in the United States and Europe.

DETAILED DESCRIPTION:
This study will evaluate the intracellular PK of TFV-DP and FTC-TP in Ghanaian HIV-infected adolescents with and without TB coinfection. As the clinical effects of TDF and FTC are related to the intracellular concentrations of the phosphate anabolites, called TFV-DP and FTC-TP, there is a need to understand the cellular pharmacology of TDF interactions in African HIV-infected adolescents with and without TB, as the study team cannot extrapolate from US patients not on antituberculosis (anti-TB) drugs. This study will enroll HIV-infected adolescents aged 10 to 18 years old with and without TB coinfection who are already established on ART. The study team hypothesize that younger age, adenosine triphosphate (ATP)-binding cassette subfamily C (ABCC) single nucleotide polymorphisms (SNPs) and anti-TB therapy may influence the intracellular TFV-DP and FTC-TP concentrations in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adolescents aged 10 to 19 years old who are stable on antiretroviral regimen containing TDF/FTC (300/200 mg daily) for at least 8 weeks.

Exclusion Criteria:

* Unable to obtain informed signed consent from parent(s) or legal guardian.
* Pregnant or breast feeding.
* Require therapy for other opportunistic infections other than tuberculosis (TB).

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents aged 10-19 years with HIV with or without TB co-infection.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Average concentration (Cav) of intracellular TFV-DP and FTC-TP in Ghanaian HIV-infected adolescents. | After at least 8 weeks of HIV therapy.
  Mean and median Cav of intracellular TFV-DP and FTC-TP in Ghanaian HIV-infected adolescents.
Area under the time-concentration curve 0-24 hours (AUC0-24h) of intracellular TFV-DP and FTC-TP in Ghanaian HIV-infected adolescents. | After at least 8 weeks of HIV therapy.
  Mean and median AUC0-24h of intracellular TFV-DP and FTC-TP in Ghanaian HIV-infected adolescents.
Cav of TFV-DP and FTC-TP PK in HIV-infected adolescents with and without TB coinfection. | After at least 8 weeks of HIV therapy.
  Geometric mean intracellular TFV-DP and FTC-TP Cav in adolescents with TB/HIV coinfection compared to those only HIV infection.
AUC0-24h of TFV-DP and FTC-TP PK in HIV-infected adolescents with and without TB coinfection. | After at least 8 weeks of HIV therapy.
  Geometric mean of intracellular TFV-DP and FTC-TP AUC0-24h in adolescents with TB/HIV coinfection compared to those with only HIV infection.

SECONDARY OUTCOMES:
Effect of age on TFV-DP and FTC-TP Cav. | After at least 8 weeks of HIV therapy.
  Geometric mean of intracellular TFV-DP and FTC-TP Cav in adolescents aged 10 - 14 years old compared to that in adolescents aged 15 - 19 years old.
Effect of age on TFV-DP and FTC-TP AUC0-24h . | After at least 8 weeks of HIV therapy.
  Geometric mean of intracellular TFV-DP and FTC-TP AUC0-24h in adolescents aged 10 - 14 years old compared to that in adolescents aged 15 - 19 years old.
Intracellular TFV-DP and FTC-TP Cav in adolescents compared to that in historical adult controls. | After at least 8 weeks of HIV therapy.
  Geometric mean of intracellular TFV-DP and FTC-TP Cav in Ghanaian HIV-infected adolescent compared to published values in adults treated with similar dosage.
Intracellular TFV-DP and FTC-TP AUC0-24h in adolescents compared to that in historical adult controls. | After at least 8 weeks of HIV therapy.
  Geometric mean of intracellular TFV-DP and FTC-TP AUC0-24h in Ghanaian HIV-infected adolescent compared to published values in adults treated with similar dosage.
Relationship between Adenosine triphosphate (ATP)-binding cassette subfamily C, member 2 (ABCC2), member 4 (ABCC4) and member 10 (ABCC10) SNPs and TFV-DP and FTC-TP AUC0-24h. | After at least 8 weeks of HIV therapy.
  Relationship between ABCC2, ABCC4 and ABCC10 SNPs and intracellular TFV-DP and FTC-TP AUC0-24h.
Prevalence and covariates of intracellular TFV-DP Cav < 95 fmol/106 cells in adolescents. | After at least 8 weeks of HIV therapy.
  Proportion of Ghanaian adolescents and factors associated with intracellular TFV-DP average concentration < 95 fmol/106 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Awewura Kwara, MD, Principal Investigator — University of Florida
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Undecided